CLINICAL TRIAL: NCT04363398
Title: Prevention of Patellar and Achilles Tendinopathies in Youth Basketball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport Injury Prevention Research Centre (Other)
Collaborators: General Electric (Industry); National Basketball Association (Unknown)
Responsible Party: Principal Investigator, Carolyn Emery, Professor, Sport Injury Prevention Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB16-0864
Record Dates: First submitted 2018-04-27; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Injury, Knee; Injury, Ankle; Tendinopathy; Sports Injuries in Children
MeSH Terms: conditions — Knee Injuries; Ankle Injuries; Tendinopathy

STUDY DESIGN:
Intervention Model Description: A Hybrid (effectiveness-implementation) Type 2 RCT design will be conducted. Teams will be randomized into either a comprehensive or standard intervention delivery group.
Who Masked: Participant, Investigator
Masking Description: Participants (teachers and students) are not aware of what arm they are randomized to. The primary investigators performing the analysis and overseeing all decisions are blinded to the schools receiving the comprehensive vs standard follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive (Experimental): Coaches from schools randomized to the comprehensive follow-up receive a workshop outlining a neuromuscular training program to be used as a warm-up for 10 minutes at the beginning of each basketball practice and game. Throughout the season, a trained research team member will monitor the team weekly for injuries, participation, and adherence, and provide support to the school coaches regarding the warm-up.
  Interventions: Other: Comprehensive Follow-up
- Standard (Active Comparator): Coaches from schools randomized to the standard follow-up receive a workshop outlining a neuromuscular training program to be used as a warm-up for 10 minutes at the beginning of each basketball practice and game. Throughout the season, a research team member will monitor the team weekly for injuries, participation, and adherence, however will not provide support to the school coaches regarding the warm-up.
  Interventions: Other: Standard Follow-up

INTERVENTIONS:
Other: Comprehensive Follow-up — Trained research staff members will provide weekly support to coaches on the NMT warm-up.
  Arms: Comprehensive
Other: Standard Follow-up — Research staff will monitor teams weekly, however no additional support for warm-up will be provided.
  Arms: Standard

SUMMARY:
This study seeks to determine the prevalence of knee and ankle tendinopathies in youth basketball players, as well as determine the efficacy of a Basketball specific Neuromuscular training warm-up in reducing injuries.

DETAILED DESCRIPTION:
1. BACKGROUND & RATIONALE Basketball is one of the most popular youth sports in the United States and Canada. Knee and ankle injuries are the most common injuries in youth basketball (40%). Patellar and Achilles tendinopathies (PATs) are of particular concern in elite level basketball with a prevalence of 32% for patellar tendinopathy in elite male athletes (60% career prevalence). The risk for injury may be initiated in youth basketball where overuse injury incidence increases with age. Previously reported PAT injury rates likely underestimate the burden of overuse injury in youth basketball as current surveillance guidelines are optimized for acute injury and there are no guidelines on appropriate tendinopathy diagnosis in youth athletes. Current knowledge on basketball-related injuries (acute and overuse) in adolescent athletic community is sparse. Jump loads, landing mechanics, joint morphology and tendon structure changes may be predictive of tendinopathy. However, their consequences on PAT risk in basketball remain to be investigated using prospective cohort study methodologies. Encouragingly, the potential for mediating injury risk in youth sport through neuromuscular training programs has been demonstrated. A basketball specific neuromuscular training program (BSpecNMT) in turn may be efficacious for primary PAT prevention. Clearly, there is an urgent need to advance the current state of injury surveillance, prevention programs, sport-specific risk factors for PATs and structural consequences of PATs in youth basketball.
2. RESEARCH OBJECTIVES Primary Objectives 1) To quantify the prevalence and severity of patellar and Achilles tendinopathies and assess associated risk factors in youth basketball (Year 1); and 2) To evaluate the efficacy of a BSpecNMT program in reducing patellar and Achilles tendinopathies and all injuries in youth basketball players (Year 2 and 3).
3. METHODS A Hybrid (effectiveness-implementation) Type 2 RCT design will be conducted. Teams will be randomized into either a comprehensive or standard intervention delivery group. All coaches will attend one pre-season coach workshop for the basketball specific neuromuscular (BSpecNMT) warm-up program. The workshop was led by a physiotherapist, athletic trainer, or strength and conditioning coach before the start of the season. During the pre-season coach workshop, coaches will take part in a theoretical and practical session about basketball injury prevention and warm-up exercises. Coaches in the both study groups will be instructed to carry out the 10-minute warm-up program at the beginning of all training sessions.

In addition, the comprehensive intervention group will receive weekly visits at team practices from a research physiotherapist, athletic trainer, or strength and conditioning coach. These visits will provide the team guidance with the BSpecNMT warm-up to facilitate proper technique and appropriate progression of the BSpecNMT warm-up exercises.

All teams will have their adherence to the BSpecNMT recorded on a weekly basis by a Team Designate. In addition, injuries will be prospectively monitored through a weekly self-report questionnaire, a post-season questionnaire (completed by players) and injury report form (completed by team designates). Also, Coaches' knowledge and attitudes to injury prevention will be registered by surveys during the pre-season, post-workshop, post-season, 6-month post-season, and 12-month post-season timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Plays competitive basketball with School or club

Exclusion Criteria:

* Injured at baseline

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 441 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Basketball injuries | Medical attention injuries daily, additional injuries weekly and a post-season interview at 4 months if needed.
  To effectively capture all injuries (i.e., acute and overuse/chronic injuries), an "all-complaint" injury definition will be adopted through year 1 and year 2 of study. An injury is any physical complaint, including any pain, ache, joint instability, stiffness or any other complaint resulting from participating in basketball-related sessions, including but irrespective of the need for medical attention (seeking care from a trainer or medical practitioner) or time-loss (inability to complete a basketball-related session, or participate in one or more days after the onset of injury) from basketball-related activities. Further, an injury is identified as acute if its onset was sudden and clearly associated with an identifiable event and overuse if its onset, whether gradual or sudden, was unidentifiable with any event.
Weekly Exposure Sheet (WES) | This will be recorded weekly during the basketball season (average 4 months)
  The duration of time players are exposed to basketball, and the basketball NMT program, will be captured. This will be captured using a previously validated Weekly Exposure Form (WES). This includes start and end time of sport sessions, attendance at those sessions, and reason for non-attendance.

SECONDARY OUTCOMES:
Player Questionnaire | This measure will be assess at baseline (pre-season) and end of the basketball season (average 4 months after baseline)
  Injury history, demographics, medical history
Coach Beliefs/Behaviors | The questionnaire will be administered to team coaches at 4 different time-points - Pre-workshop at baseline, post workshop at baseline, post-season at 4 months, post-season follow-up at 6 months and post-season follow-up at 12 months.
  Coach knowledge, experiences, attitudes and beliefs of the coach related to injury prevention and the neuromuscular training program will be assessed through a previously validated Health Action Process Approach questionnaire adapted in previous studies in a similar setting

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Emery, PT, PhD, Principal Investigator — Sport Injury Prevention Research Centre, University of Calgary
Locations (1):
- Sport Injury Prevention Research Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No